CLINICAL TRIAL: NCT01156415
Title: A 52-week, Multi-center, Open-label Study of the Safety and Tolerability of Agomelatine Sublingual Tablets in Patients With Major Depressive Disorder (MDD)
Brief Title: Open-label Long Term (52 Weeks) Safety and Tolerability of Agomelatine Sublingual Tablets in Major Depressive Disorder (MDD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAGO178C2399
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2013-03

CONDITIONS: Major Depressive Disorder
Keywords: agomelatine; Major Depressive Disorder; MDD; depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — agomelatine

ARMS (2):
- Agomelatine (AGO178) 0.5 mg (Experimental)
  Interventions: Drug: AGO178
- Agomelatine (AGO178) 1 mg (Experimental)
  Interventions: Drug: AGO178

INTERVENTIONS:
Drug: AGO178
  Arms: Agomelatine (AGO178) 1 mg
Drug: AGO178
  Arms: Agomelatine (AGO178) 0.5 mg

SUMMARY:
The study will assess safety and tolerability of 0.5 mg/day and 1 mg/day of sublingual (under the tongue) formulation of agomelatine (AGO178) in patients with Major Depressive Disorder over a 52-week open-label phase.

Cohort I is restricted to include patients who have completed a previous Novartis agomelatine (178C) Double-blind study.

Cohort II will include de-novo patients (those who did not participate in a previous agomelatine 178C study) and will only be open for a limited time span ranging from approximately June to Sept 2010, at which point this cohort II will be closed to enrollment.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria Cohort I:

* Documentation of completion of a Novartis AGO178C Double-blind Study in MDD patients.
* Male and female adults, 18 through 71 years of age, inclusive (i.e., same age range as for Double-blind Study, but with upper age limit increased by 1-year to accommodate patients whose age increased during the Double-blind Study).
* Female patients should continue to use effective contraception as defined in double-blind study protocol.

Inclusion Criteria:

Key Inclusion criteria Cohort II:

* Male and female adults, 18 through 70 years of age, inclusive.
* Diagnosis of MDD, single or recurrent episode, according to DSM-IV criteria.
* Current episode ≥4 weeks.
* CGI-Severity score ≥4 at Screening and Baseline.

Exclusion Criteria:

Key Exclusion Criteria Cohort I:

* Concomitant use of fluvoxamine.
* Any significant medical condition that emerged during Double-blind Phase of a previous study, which may interfere with study participation and/or study assessments as assessed by the investigator.

Exclusion Criteria:

Key Exclusion criteria Cohort II:

* History of bipolar disorder (I or II), schizophrenia, schizoaffective disorder, eating disorder (current or during previous one year), obsessive-compulsive disorder.
* Any other current Axis I disorder other than MDD which is the focus of treatment.
* Substance or alcohol abuse in the last 30 days, dependence in the last 6 months.
* Prior exposure to agomelatine.
* Female patients of childbearing potential who are not using effective contraception.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 837 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Reports of adverse events, serious adverse events, changes in laboratory values, ECGs, vital signs, physical examination, and Columbia Suicidality Severity Rating Scale | 52 weeks

SECONDARY OUTCOMES:
Change from Baseline to Week 6, 8, 12, 28, 36 and 52 on total score of the Hamilton Depression Rating Scale | Week 6, 8, 12, 28, 36 and 52
Proportion of patients who demonstrate clinical improvement at Week 6,8,12, 28,36 and 52, where improvement is defined by a score of 1 or 2 on the CGI-I scale | Week 6, 8, 12, 28, 36 and 52
Overall illness severity as measured by change from Baseline on CGI-S (Clinical Global Impression of severity scale) at week 52 | Week 52
Patients' ability to function in daily life as measured by change from Baseline on total score of Sheehan Disability Scale at week 52 | Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (98):
- United States (95):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Advanced Research Associates, Glendale, Arizona
  - Southwest Health Ltd dba The Mollen Clinic, Scottsdale, Arizona
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Southwestern Research Institute, Beverly Hills, California
  - Comprehensive Neuroscience, Cerritos, California
  - ATP Clinical Research, Inc, Costa Mesa, California
  - Collaborative Neuroscience Network, Garden Grove, California
  - Pharmacology Research Institute, Newport Beach, California
  - Pacific Clinical Research Medical Group, Orange, California
  - CNRI-San Diego, LLC, San Diego, California
  - University of California, San Diego Medical Center, San Diego, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Viking Clinical Research Center, Temecula, California
  - Collaborative Neuroscience, Torrance, California
  - University of Colorado, Aurora, Colorado
  - Western Affiliated Research Institute, Denver, Colorado
  - Middlesex Hospital, Middletown, Connecticut
  - Clinical Studies, Altamonte Springs, Florida
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Arocha Research Center, Coral Gables, Florida
  - CNS Clinical Research, Coral Springs, Florida
  - Sjs Clinical Research, Destin, Florida
  - MD Clinical, Hallandale, Florida
  - CNS Healthcare, Jacksonville, Florida
  - Florida Clinical Research Center, Maitland, Florida
  - CNS Healthcare, Orlando, Florida
  - Quantum Lab. at N. Broward Memory Disorder Center, Pompano Beach, Florida
  - Miami Research Associates, South Miami, Florida
  - Comprehensive NeuroScience, Inc., St. Petersburg, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Hawaii Clinical Research Center, Honolulu, Hawaii
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Joliet Center for Clinical Research, Joliet, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - Rush University Medical Center, Skokie, Illinois
  - Deaconess Clinic Gateway, Newburgh, Indiana
  - Pharmasite Research, Pikesville, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Mount Auburn Medical Associates, Watertown, Massachusetts
  - Coastal Research Associates, Weymouth, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - Pine Rest Christian Mental Health Services, Grand Rapids, Michigan
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Comprehensive Psychiatric Associates, Gladstone, Missouri
  - Robert Wood Johnson Medical School, Piscataway, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - CRI Worldwide, Willingboro, New Jersey
  - Albuquerque Neuroscience, Albuquerque, New Mexico
  - Neurological Associates Of Albany, Albany, New York
  - Social Psychiatry Research, Inc./ SPRI, Brooklyn, New York
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Eastside Comprehensive Medical Service, New York, New York
  - Medical & Behavior Health Research, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Montefiore Medical Center, The Bronx, New York
  - Pharmquest, Greensboro, North Carolina
  - Zarzar Psychiatric Associates, Raleigh, North Carolina
  - Piedmont Medical Research Associates, Inc., Winston-Salem, North Carolina
  - Odyssey Research Services, Fargo, North Dakota
  - Neuro Behavioral Clinical Research, Canton, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - North Star Medical Research, Cleveland, Ohio
  - The Ohio State Universtiy - Harding Hospital, Columbus, Ohio
  - Neurology & Neuroscience Center of Ohio, Toledo, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - SP Research, Oklahoma City, Oklahoma
  - Cutting Edge Research, Oklahoma City, Oklahoma
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Oregon Center for Clinical Investigations, Portland, Oregon
  - Summit Research, Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Research Strategies of Memphis, Memphis, Tennessee
  - Clinical Research Associates, Nashville, Tennessee
  - Millwood Hospital, Arlington, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Bayou City Research Limited, Houston, Texas
  - Claghorn Lesem Research Clinic, Inc., Houston, Texas
  - Texas Center for Drug Development, Houston, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Radiant Research, Salt Lake City, Utah
  - University of Utah Mood Disorders Clinic, Salt Lake City, Utah
  - Alliance Research Group, LLC, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Frontier Institute, Spokane, Washington
  - Independent Psychiatric Consultants, Waukesha, Wisconsin
- Puerto Rico (3):
  - Centro de Investigacion Clinica Psiquiatrica, Ponce
  - Dharma Institute and Research Center, San Juan
  - INSPIRA Clinical Research, San Juan

REFERENCES:
- See also: Results for CAGO178C2399 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=7243